CLINICAL TRIAL: NCT04237506
Title: Targeted Ballet Class for Increased Range of Motion and Stretch Reflex Regulation in Cerebral Palsy
Brief Title: Targeted Ballet Class for Cerebral Palsy
Acronym: TBCCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Citlali Lopez-Ortiz (Other)
Responsible Party: Sponsor-Investigator, Citlali Lopez-Ortiz, Principal Investigator, University of Illinois at Urbana-Champaign
Organization: University of Illinois at Urbana-Champaign (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16718; 16CN1335 (Other: Carle Foundation Hospital IRB, Urbana IL)
Record Dates: First submitted 2019-12-31; First posted 2020-01-23 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Children and adults with cerebral palsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): All participants in this group will take the one-hour ballet dance class twice per week for six weeks
  Interventions: Behavioral: Targeted ballet dance

INTERVENTIONS:
Behavioral: Targeted ballet dance — The one-hour ballet dance class will be provided twice per week for six weeks. The syllabi are adapted from the Joffrey Ballet Academy and Royal Academy of Dancing that are targeting grades primary to level 1 and typically developing kids at the age of 6 to 10 years old. PI will be the class instructor, and the class structure will follow the guidelines in 'Dance program for physical rehabilitation and participation in children with cerebral palsy' by Lopez-Ortiz et al.

SUMMARY:
This study aims to investigate the effect of the targeted ballet dance on participants with cerebral palsy

DETAILED DESCRIPTION:
Cerebral palsy (CP) is the most common motor disorder in childhood, with a prevalence of 3.1 to 3.6 cases per 1000 living births in the United States. The motor signs of CP include abnormal muscle tone and motor control, preventing individuals with CP from participating in normal daily activity. The most common type of CP is spastic CP, in which spasticity is present and range of motion in the joints is reduced. Physical therapy is one fundamental method of rehabilitation that attempts to recover motor function via exercises, while the effects of physical therapy are still elusive due to the lack of comprehensive evidence. This study uses a targeted ballet class to promote balance, increased range of motion, and reduced spasticity. The combination of qualitative clinical measures and quantitative assessment spasticity aims to demonstrate the benefits brought by the dance class.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with spastic cerebral palsy
* is between 3 to 64 years old
* have no uncorrected vision
* have no other neuromuscular or musculoskeletal condition
* have not had surgical procedures within six months of enrollment in the study
* participate in stable school and/or private physical therapy with a frequency no greater than one session per week
* have no changes in medication for the last six months
* have the ability to pay attention and follow three-step directions
* be medically stable, (8) have no other concurrent illness
* have not received any Botox treatment within three months previous to the initiation of the study, and have Gross Motor System Classification Scale (GMFCS) I-IV (NOT V).

Exclusion Criteria:

* Not meeting ALL of the criteria

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2021-02-13 (Actual)

PRIMARY OUTCOMES:
Change in Montreal Stretch Reflex Threshold | Tested during assessment sessions and on the first and last week of dance to evaluate change from the baseline at a 10-week period.
  Montreal Stretch Reflex threshold is an objective method using surface electromyography and electrogoniometer to quantify spasticity by measuring the onset of the tonic stretch reflex.

SECONDARY OUTCOMES:
Change in Selective control assessment of the lower extremity (SCALE) Score Sheet | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  Selective control assessment of the lower extremity (SCALE) evaluates the ability to perform isolated movements at one joint without activation of other joints or flexor/extensor patterns. It has been shown to have high interrater reliability. SCALE scores the isolated movement at five joints of one lower limb, including hip, knee, foot/subtalar joint, ankle and toe. For each joint, the movement is rated on a scale of 0 to 2 that a score of 0 indicates inability to perform the action and a score of 2 indicates normal movement. The scores are summed to obtain a total score for that limb (the maximum score is 10), and a high score indicates a better capacity of selectively controlling movements of the joint.
Change in Pediatric Berg Balance Scale (PBS) | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  It assesses balance function in children and has been shown to have good reliability and validity. It has 14 items and each item is scored on a scale of 0 to 4 that a score of 4 indicates the ability to perform the task with minimal or no assistance. The total score is obtained by adding individual scores of each item together, and a higher score indicates better balance function.
Change in Dyskinesia impairment scale (DIS) | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  It has two subscales, dystonia and choreoathetosis, and is used to assess the severity of dystonia and choreoathetosis during activity or rest. It has been shown to have good to excellent reliability and validity. In each subscale, the score is rated on a scale of 0 to 4 for both duration and amplitude of each criterion that a score of 0 indicate normal movement and a score of 4 indicates that the motor symptom is always present. The scores will be added together to obtain two subscores, and the total score is the sum of subscores (the highest possible score is 576) and the higher the total score is, the more severs the dystonia or choreoathetosis will be.
Participant Information Questionnaire | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  Questionnaire on health status and demographic information
Change in Quality fo Upper Extremity Skills Test (QUEST) | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  It has 36 items that evaluate the upper and hand functions with excellent test reliability. The score of each item ranges from -1 to 2. A score of 2 indicates the ability to complete actions as requested, a score of 1 indicate being unable or unwilling to complete actions, or unable to administer the item. A score of -1 is given when abnormal movement is present in the posture section. Initial scores are obtained by adding scores from each section, and these initial scores is standardized to get the total score which ranges from 0 to 100. The higher the score, the better upper limb function will be.
Change in Gross Motor Function Classification Scale | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  It evaluates gross motor function with 5 levels with level 5 being the most impaired that requires assistance at all settings (at home, school, outdoors and in the community).
Change in Modified Tardieu Scale | Tested during assessment sessions to measure change from the baseline at a 10-week period.
  It evaluates spasticity by measuring the angle of catch and range of motion. Angle of catch is the joint angle at which there is a resistance of muscle when it is passively stretched at different speeds, and range of motion is the range a joint can achieve when the muscle is stretched at a very slow speed. Scores range from 0 to 5. A score of 0 means no resistance of the muscle during the passive movement and a score of 5 indicate the joint immobility.

CONTACTS AND LOCATIONS:
Overall Officials: Citlali López-Ortiz, M.A., Ph.D, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

REFERENCES:
- [Background] Lopez-Ortiz C, Gladden K, Deon L, Schmidt J, Girolami G, Gaebler-Spira D. Dance program for physical rehabilitation and participation in children with cerebral palsy. Arts Health. 2012 Feb 1;4(1):39-54. doi: 10.1080/17533015.2011.564193. Epub 2011 Jun 13. PMID 25431617
- [Background] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Background] Rodrigues, Marcos & Levin, Mindy & Feldman, Anatol & Mullick, Aditi. (2014). A New Standard in Objective Measurement of Spasticity. Journal of Medical Devices. 7. 10.1115/1.4024488.
- [Background] Lopez-Ortiz C, Gaebler-Spira DJ, Mckeeman SN, Mcnish RN, Green D. Dance and rehabilitation in cerebral palsy: a systematic search and review. Dev Med Child Neurol. 2019 Apr;61(4):393-398. doi: 10.1111/dmcn.14064. Epub 2018 Oct 23. PMID 30350851
- [Background] Chen CL, Shen IH, Chen CY, Wu CY, Liu WY, Chung CY. Validity, responsiveness, minimal detectable change, and minimal clinically important change of Pediatric Balance Scale in children with cerebral palsy. Res Dev Disabil. 2013 Mar;34(3):916-22. doi: 10.1016/j.ridd.2012.11.006. Epub 2013 Jan 3. PMID 23291508
- [Background] Lopez-Ortiz C, Egan T, Gaebler-Spira DJ. Pilot study of a targeted dance class for physical rehabilitation in children with cerebral palsy. SAGE Open Med. 2016 Sep 23;4:2050312116670926. doi: 10.1177/2050312116670926. eCollection 2016. PMID 27721977
- [Background] Gracies JM, Burke K, Clegg NJ, Browne R, Rushing C, Fehlings D, Matthews D, Tilton A, Delgado MR. Reliability of the Tardieu Scale for assessing spasticity in children with cerebral palsy. Arch Phys Med Rehabil. 2010 Mar;91(3):421-8. doi: 10.1016/j.apmr.2009.11.017. PMID 20298834
- [Background] Klingels K, De Cock P, Desloovere K, Huenaerts C, Molenaers G, Van Nuland I, Huysmans A, Feys H. Comparison of the Melbourne Assessment of Unilateral Upper Limb Function and the Quality of Upper Extremity Skills Test in hemiplegic CP. Dev Med Child Neurol. 2008 Dec;50(12):904-9. doi: 10.1111/j.1469-8749.2008.03123.x. Epub 2008 Sep 20. PMID 18811701
- [Background] Graham HK, Rosenbaum P, Paneth N, Dan B, Lin JP, Damiano DL, Becher JG, Gaebler-Spira D, Colver A, Reddihough DS, Crompton KE, Lieber RL. Cerebral palsy. Nat Rev Dis Primers. 2016 Jan 7;2:15082. doi: 10.1038/nrdp.2015.82. PMID 27188686
- [Derived] Lopez-Ortiz C, He M, Gaebler-Spira D, Levin MF. Learning ballet technique modulates the stretch reflex in students with cerebral palsy: case series. BMC Neurosci. 2024 Nov 6;25(1):66. doi: 10.1186/s12868-024-00873-0. PMID 39506647